CLINICAL TRIAL: NCT05948657
Title: ESCAPE - Evaluation of Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography in Active Surveillance for Prostate CancEr
Brief Title: Evaluation of Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography in Active Surveillance for Prostate CancEr
Acronym: ESCAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-03025893
Record Dates: First submitted 2023-06-20; First posted 2023-07-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will undergo PSMA-PET CT (Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography) at baseline, 12 month and 24 month time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PSMA-PET CT (Other): Patients will undergo PSMA-PET CT (Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography) at baseline, 12 month and 24 month time point.
  Interventions: Diagnostic Test: PSMA-PET CT

INTERVENTIONS:
Diagnostic Test: PSMA-PET CT — Patients will undergo PSMA-PET CT (Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography) at baseline, 12 month and 24 month time point.

SUMMARY:
This study will be assessing the ability of PSMA-PET CT to determine the absence of clinically significant prostate cancer in patients on active surveillance (AS) with low risk and favorable intermediate-risk prostate cancer.

DETAILED DESCRIPTION:
This is a prospective, multicenter, nonrandomized single-arm study assessing the diagnostic accuracy of PSMA-PET CT (Prostate Specific Membrane Antigen Positron Emission Tomography-Computed Tomography) in determining the absence of clinically significant prostate cancer in patients on active surveillance (AS).The trial will enroll 200 subjects for low and favorable intermediate-risk prostate cancer patients per NCCN guidelines who have elected to pursue active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥ 18.
* Histologically confirmed low or favorable intermediate risk prostate cancer per NCCN guidelines. (Note: Grade Group 2 must have 20% or less involvement in every core and no presence of cribiform or intraductal carcinoma).
* PSA < 20 ng/ml.
* Ability to undergo yearly PSMA-PET CT.
* Ability to undergo yearly prostate mpMRI.
* Ability to undergo transrectal or transperineal template and fusion prostate biopsy.
* Ability to complete HRQOL surveys (EPIC, IPSS, IIEF-5).
* Willingness to undergo yearly prostate biopsies.

Exclusion Criteria:

* History of prior treatment for prostate cancer.
* History of systemic therapy for prostate cancer.
* Inability to undergo transrectal ultrasound.
* Life expectancy less than 10 years.
* Not interested in pursuing active surveillance.
* Initial diagnosis of prostate cancer greater than 15 months.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) | Baseline
  Negative predictive value (NPV): The NPV is defined as the number of negative image results with identified clinically insignificant prostate cancer on biopsy divided by the number of negative image results.
Negative predictive value (NPV) | 12 months
  Negative predictive value (NPV): The NPV is defined as the number of negative image results with identified clinically insignificant prostate cancer on biopsy divided by the number of negative image results.
Negative predictive value (NPV) | 24 months
  Negative predictive value (NPV): The NPV is defined as the number of negative image results with identified clinically insignificant prostate cancer on biopsy divided by the number of negative image results.

SECONDARY OUTCOMES:
Positive predictive value (PPV) of PSMA PET. | Baseline
  PPV of PSMA PET. Positive predictive value (PPV): The PPV is defined as the number of positive image results with identified csPCa on biopsy divided by the number of positive image results.
Positive predictive value (PPV) of PSMA PET. | 12 months
  PPV of PSMA PET. Positive predictive value (PPV): The PPV is defined as the number of positive image results with identified csPCa on biopsy divided by the number of positive image results.
Positive predictive value (PPV) of PSMA PET. | 24 months
  PPV of PSMA PET. Positive predictive value (PPV): The PPV is defined as the number of positive image results with identified csPCa on biopsy divided by the number of positive image results.
Number of patients with negative PSMA pet scan. | Baseline
Number of patients with negative PSMA pet scan. | 12 months
Number of patients with negative PSMA pet scan. | 24 months
Number of positive scans on mpMRI | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on mpMRI | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on mpMRI | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on PSMA-PET | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on PSMA-PET | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on PSMA-PET | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on both PSMA-PET and mpMRI | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on both PSMA-PET and mpMRI | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of positive scans on both PSMA-PET and mpMRI | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Sensitivity: The sensitivity will be defined as the number of positive image results with a csPCa upon biopsy divided by the number of biopsied patients with csPCa following the imaging.
Number of negative scans on mpMRI | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on mpMRI | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on mpMRI | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on PSMA-PET | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on PSMA-PET | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on PSMA-PET | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on both PSMA-PET and mpMRI | Baseline
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on both PSMA-PET and mpMRI | 12 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of negative scans on both PSMA-PET and mpMRI | 24 months
  Specificity and sensitivity of PSMA-PET, mpMRI, and the combination.
  Specificity: The specificity is defined as the number of negative image results followed by the absence of csPCa in the corresponding biopsy divided by the number of biopsies that did not identify csPCa.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by PSMA-PET. | Baseline
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by PSMA-PET. | 12 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by PSMA-PET. | 24 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by mpMRI. | Baseline
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by mpMRI. | 12 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected by mpMRI. | 24 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected on PSMA-PET and mpMRI. | Baseline
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected on PSMA-PET and mpMRI. | 12 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.
Number of patients who have clinically significant Prostate Cancer (csPCa) detected on PSMA-PET and mpMRI. | 24 months
  The proportion of csPCa detected by PSMA-PET, mpMRI, and the combination. Proportion of patients with csPCa: this will be the number of patients identified as having csPCa divided by the number of patients with a biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy McClure, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - Case Western University Hospitals, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No